CLINICAL TRIAL: NCT07277894
Title: The Effect of Virtual Reality During Non-Invasive Urodynamics on Patients' Vital Signs, Anxiety, and Satisfaction Levels
Brief Title: The Effect of Virtual Reality During Urodynamics on Vital Signs, Anxiety, and Satisfaction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Esra Özden, Principal Investigator and Lecturer, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SagligBilimleriU
Record Dates: First submitted 2025-08-22; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Urinary Incontinence; Urodynamic Studies; Urodynamics
Keywords: Urinary incontinence; urodynamic studies; anxiety; satisfaction
MeSH Terms: conditions — Urinary Incontinence; Anxiety Disorders; Personal Satisfaction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- virtual reality group (Experimental): In the course of noninvasive urodynamic testing, patients will be presented with a 360-degree visualization of a clean and spacious bathroom environment via virtual reality goggles.
  Interventions: Other: Virtual reality group
- Control group (No Intervention): The control group participants will not be equipped with virtual reality headsets, and only routine clinical procedures will be administered.

INTERVENTIONS:
Other: Virtual reality group — In the course of noninvasive urodynamic testing, patients will be presented with a 360-degree visualization of a clean and spacious bathroom environment via virtual reality goggles.
  Arms: virtual reality group

SUMMARY:
Study Topic

This research aims to evaluate the effects of virtual reality (VR) application during noninvasive urodynamics on patients' vital signs, anxiety, and satisfaction levels.

Significance of the Problem

Urodynamic studies are essential diagnostic methods for assessing lower urinary tract functions.

However, they often cause discomfort, pain, and high levels of anxiety in patients.

This not only negatively affects the patient experience but also creates uncertainty in clinical decision-making.

Previous studies have shown that nursing interventions such as music therapy, aromatherapy, and heating pads effectively reduce anxiety.

Recently, VR technology has emerged as a promising tool to distract patients, thereby reducing pain and anxiety.

Aim of the Study

To investigate the effects of VR application during noninvasive urodynamics on:

Vital signs,

Anxiety,

Comfort, and

Patient satisfaction.

Methodology

Design: Single-center, randomized controlled clinical trial.

Setting/Duration: Urology Outpatient Clinic, Ankara Etlik City Hospital, September - December 2025.

Sample: Based on power analysis, at least 26 patients per group; total minimum of 52 participants.

Inclusion criteria: 18-50 years old, undergoing noninvasive urodynamics for the first time, voluntary participation.

Exclusion criteria: Previous urodynamics, use of anxiolytics/antidepressants, communication/vision/balance impairments.

Randomization: Block randomization (block size 6).

Data Collection Tools

Descriptive Characteristics Form

State-Trait Anxiety Inventory (STAI)

Vital Signs and Urodynamic Parameters Monitoring Form

Patient Satisfaction and Comfort Assessment (Visual Analog Scale - VAS)

VR Application Satisfaction Form

Interventions

VR Group: During uroflowmetry, patients will experience a 360° virtual hygienic and spacious bathroom environment via VR goggles.

Control Group: Routine clinical practice only, with standard pre-procedure information.

Data Analysis

Data will be analyzed using SPSS 21.0.

Normality will be tested with Kolmogorov-Smirnov.

Between-group differences will be assessed using Independent Samples t-test or Mann-Whitney U test, as appropriate.

Statistical significance will be set at p < 0.05.

Ethical Considerations

Ethical approval and hospital permission were obtained.

Informed consent will be collected from all participants prior to data collection.

DETAILED DESCRIPTION:
Background:

Urodynamic studies are essential diagnostic tools for evaluating lower urinary tract function. However, they often cause discomfort, pain, and anxiety, which may negatively affect patient experience and the accuracy of clinical results. Non-pharmacological interventions such as music therapy and aromatherapy have been shown to reduce anxiety. Virtual reality (VR) is a promising new approach that provides immersive distraction and has demonstrated benefits in clinical care, but its use in urodynamic testing remains limited.

Objective:

To evaluate the effects of VR application during non-invasive urodynamics on:

Vital signs

Anxiety

Comfort

Patient satisfaction

Design and Setting:

Single-center, randomized controlled clinical trial. Location: Urology Outpatient Clinic, Ankara Etlik City Hospital. Study period: November 2025 - January 2026.

Participants:

Minimum 52 participants (26 per group).

Inclusion criteria: Adults aged 18-50, undergoing non-invasive urodynamics for the first time, voluntary participation.

Exclusion criteria: Previous urodynamics, antidepressant/anxiolytic use, communication problems, visual or balance disorders.

Randomization:

Block randomization (block size = 6).

Interventions:

VR Group: During uroflowmetry, participants will use VR goggles displaying a 360° visualization of a hygienic and spacious bathroom environment.

Control Group: Routine clinical practice only, with standard pre-procedure information.

Measurements and Tools:

Descriptive Characteristics Form

State-Trait Anxiety Inventory (STAI)

Vital Signs and Urodynamic Parameters Monitoring Form

Patient Satisfaction and Comfort Assessment (Visual Analog Scale, VAS)

VR Application Satisfaction Form

Data Collection and Analysis:

Assessments conducted before, during, and after urodynamics.

Statistical analyses with SPSS 21.0.

Normality tested with Kolmogorov-Smirnov.

Group comparisons with Independent Samples t-test or Mann-Whitney U test.

Significance level: p < 0.05.

Ethics:

Approved by the Gülhane Research Ethics Committee. Institutional approval obtained. Written informed consent will be collected from all participants.

Expected Contribution:

This trial will provide evidence on the role of VR in reducing anxiety, improving comfort, and enhancing patient satisfaction during urodynamic procedures.

ELIGIBILITY:
Inclusion Criteria:

* Being the first to undergo noninvasive urodynamics;
* Agreeing to participate in the study;
* Being between the ages of 30-50.

Exclusion Criteria:

* Having had a urodynamic test before;
* Being on antidepressants or anxiolytics;
* Having communication and cooperation problems;
* Having visual or balance disorders.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Change in State Anxiety Score (State-Trait Anxiety Inventory - STAI-State) | Baseline and immediately after the procedure
  State Anxiety will be assessed using the State-Trait Anxiety Inventory (STAI-State), a 20-item scale ranging from 20 to 80 points. Higher scores indicate higher anxiety. Unit of Measure: points (20-80)

SECONDARY OUTCOMES:
Uroflowmetry Parameters (Qmax, Qavg, voided volume, flow time) | During the procedure
  Uroflowmetry parameters including maximum flow rate (Qmax, mL/s), average flow rate (Qavg, mL/s), voided volume (mL), and flow time (seconds) will be recorded during the procedure. Unit of Measure: mL/s; mL; seconds
Change in Vital Signs (blood pressure, heart rate, respiratory rate, oxygen saturation) | Baseline and immediately after procedure
  Vital signs (systolic/diastolic blood pressure in mmHg, heart rate in bpm, respiratory rate in breaths/min, and SpO₂ in %) will be measured before and after the uroflowmetry procedure. Unit of Measure: mmHg, bpm, breaths/min, %
Patient Satisfaction Score (Visual Analog Scale - VAS) | Immediately after the procedure
  Satisfaction will be assessed using a Visual Analog Scale ranging from 0 (no satisfaction) to 10 (highest satisfaction). Unit of Measure: VAS score (0-10)
Patient Comfort Score (Visual Analog Scale - VAS) | Immediately after the procedure
  Comfort will be assessed using a Visual Analog Scale ranging from 0 (no comfort) to 10 (highest comfort). Unit of Measure: VAS score (0-10)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) related to primary and secondary outcomes will be shared. Supporting information including the study protocol, statistical analysis plan (SAP), informed consent form (ICF), and clinical study report (CSR) will also be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available beginning 6 months after publication of the primary study results and will remain accessible for up to 5 years.
Access Criteria: Access will be provided to qualified researchers who submit a methodologically sound proposal and obtain approval from an independent ethics committee. Requests should be directed to the Principal Investigator via institutional email.